CLINICAL TRIAL: NCT07087457
Title: The Effect of Human and Digital Stimulus Exercise Interventions Based on the Transtheoretical Model on Increasing Physical Activity Levels in Sedentary Office Workers: A Randomized Crossover Study
Brief Title: The Effect of Transtheoretical Model-Based Exercise Interventions on Increasing Physical Activity in Office Workers
Acronym: FIT-MOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sebahat Gozum, Proffesor, Akdeniz University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: TBAEK-164
Record Dates: First submitted 2025-06-30; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Office Workers; Sedanter
Keywords: Sedentary lifestyle; inactivity; office workers; transthoretical model; digital stimuli; physical activity; hearth rate
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A-The digital stimulus command (Experimental): The digital stimulus command:
  This group will receive only digital alerts for 4 weeks. Following the washout period, they will participate in a 5-day, 30-minute walking program, accompanied by a researcher, for 4 weeks.
  Interventions: Behavioral: The digital stimulus command; Behavioral: 5 day 30-minute walking program
- Group B- 5-day 30-minute walking program (Experimental): 5 day 30-minute walking program. This group will participate in a 30-minute walking program for 5 days a week, accompanied by a researcher, for 4 weeks. Following the washout period, they will receive in the digital stimulus commands for 4 weeks.
  Interventions: Behavioral: The digital stimulus command; Behavioral: 5 day 30-minute walking program

INTERVENTIONS:
Behavioral: The digital stimulus command — The digital stimulus command: Providing information on the harms of inactivity and sedentary lifestyle on online, digital platforms. The individual will take the HRV measurement in a sitting position for 5 minutes every morning (before consuming tobacco products for smokers) as taught and will send the screenshot of the data to the researcher via WhatsApp. Ensuring that the digital stimulus commands that will remind the activity in line with TTM are followed by reminders sent to the computer screen or mobile phones. Taking a break from sitting when the command "It's time for activity" comes (taking a total of 6 breaks in the working hours of 08:30 - 17:30, 1 every 60 minutes recording the activity as "completed" in the digital diary and survey form) *Activities of office workers other than the time they spend sitting; Recording the number of steps and activities in the office, its surroundings and in daily life in a digital diary.
Behavioral: 5 day 30-minute walking program — 5 day 30-minute walking program. This group was also defined as the human stimulus group because, in addition to the digital stimulus command, they will be invited by the researcher and will participate in the walking program with the researcher. This group will first receive the activity program and simultaneously will also receive the digital stimulus command interventions.

SUMMARY:
This study aims to evaluate the effect of human and digital stimulus exercise interventions based on the transtheoretical model on increasing physical activity levels in sedentary office workers. In the study, which is planned to be conducted with a randomized crossover design, participants will be randomly assigned to different intervention conditions (human and digital stimulus). Interventions will be structured in accordance with the behavior change stages of individuals and will be implemented over a certain period of time. Within the scope of the study, physiological indicators such as heart rate variability will be evaluated along with physical activity level. This study is aimed to contribute to the development of evidence-based intervention models to support the physical activity habits of individuals working in an office environment.

Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

* Office workers scoring <600 METdk/week according to the FAA survey Employees who agreed to participate in the study. Employees who are in reflection and preparation stages of TTM change.

Exclusion Criteria:

* Part-time workers, Pregnant women, People with health problems that may increase the risk of walking (musculoskeletal system disorders, people with advanced heart failure diagnosis (based on self-report), rheumatologic, etc.) Workers who are in not thinking, moving and sustaining stages of TTM change.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
1. Physical Activity Assessment | At baseline, in the washout period after intervention A (6th week) and after intervention B (11th week)
  International Physical Activity Questionnaire Short Form: The questionnaire consists of seven questions covering all types of physical activity. Physical activity levels are categorized as physically inactive, low physical activity, and adequate physical activity.
Transtheoretic Model Scale for physical activity | At baseline, in the washout period after intervention A (6th week) and after intervention B (11th week)
  This scale has four dimensions.
  1. Exercise Stages of Change: The scale consists of a single question with five options. Based on participants' responses, the exercise stage of change they are in is determined.
  2. Exercise Change Processes: The scale consists of 28 items, 10 sub-dimensions, and two main processes (cognitive and behavioral). Cognitive processes include increased awareness, dramatic help/emotional revitalization, environmental reappraisal, self-reappraisal, and social liberation. Behavioral processes include contrast/opposition, helping relationships, reinforcement management, self-liberation, and stimulus control.
  3. Exercise Self-Efficacy: This scale aims to assess an individual's strengths regarding exercise behavior.
  4. Exercise Decision-Making Balance: Explains the cognitive factors and motivational factors that play a role in the decision-making process for the individual's exercise behavior.

SECONDARY OUTCOMES:
Heart Rate Variability | At baseline, during the washout period after intervention A (week 6), and after intervention B (week 11)
  Heart Rate Variability is an important physiological indicator related to the interactions between the sympathetic and parasympathetic divisions of the autonomic nervous system. HRV, a control system used to regulate unconscious actions such as heart function, respiration, digestion, blood pressure, urination, and pupil dilation/contraction, is used to analyze the autonomic nervous system. In our study, we will use the Polar H10 Chest Strap, a widely used research tool, to determine HRV. In a validation study, linear HRV measurements obtained from the Polar H10 chest strap demonstrated strong agreement compared to ECG recordings.